CLINICAL TRIAL: NCT00045201
Title: Phase I Trial of OSI-774 and CPT-11 in Patients With Advanced Solid Tumors
Brief Title: Erlotinib Hydrochloride and Irinotecan Hydrochloride in Treating Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00015; NCI-2009-00015 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000256910; 594-02 01; NCI-5351; MAYO-MC0112; MC0112 (Other: Mayo Clinic in Rochester); 5351 (Other: CTEP); P30CA015083 (NIH); U01CA069912 (NIH); NCT01646892 (obsolete NCT alias); NCT01664286 (obsolete NCT alias)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Adult Solid Neoplasm
MeSH Terms: interventions — Erlotinib Hydrochloride; Irinotecan

ARMS (1):
- Treatment (enzyme inhibitor, chemotherapy) (Experimental): Patients receive oral erlotinib hydrochloride daily on days -6 to -1. Patients then receive irinotecan hydrochloride IV over 90 minutes on day 1 and oral erlotinib hydrochloride once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Erlotinib Hydrochloride; Drug: Irinotecan Hydrochloride

INTERVENTIONS:
Drug: Erlotinib Hydrochloride — Given orally
  Other Names: CP 358; CP-358; Cp-358,774; CP358; OSI 774; OSI-774; OSI774; Tarceva
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; CPT11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U 101440E; U-101440E; U101440E

SUMMARY:
Phase I trial to study the effectiveness of combining erlotinib hydrochloride with irinotecan hydrochloride in treating patients who have advanced solid tumors. Erlotinib hydrochloride may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining erlotinib hydrochloride and chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of erlotinib (erlotinib hydrochloride) and irinotecan (irinotecan hydrochloride), in relation to presence or absence of UGT1A1*28 polymorphism, in patients with advanced solid tumors that overexpress epidermal growth factor receptor.

II. Determine the dose-limiting toxicity of these regimens in these patients. III. Determine whether erlotinib alters the disposition of irinotecan using a previously described limited sampling model.

IV. Determine factors that influence the disposition of these drugs, including genetic variation in UGT1A1 and BCRP, in patients treated with these regimens.

V. Determine factors that influence the disposition of these drugs, in terms of tumor BCRP-expression, in tumor samples from patients treated with these drugs at the MTD.

VI. Evaluate the effect of this regimen on epidermal growth factor receptor phosphorylation in these patients.

VII. Assess, preliminarily, any antitumor activity in patients treated with these regimens.

VIII. Correlate, preliminarily, EGFR phosphorylation and/or BCRP -expression with response in tumor samples from these patients.

OUTLINE: This is a dose-escalation study. Patients are stratified according to UGTA1A genotype (all patients regardless of genotype [closed to accrual as of 9/15/04] vs UGT1A1 6/6 genotype vs UGTA1A 6/7 or 7/7 genotype).

Patients receive oral erlotinib hydrochloride daily on days -6 to -1. Patients then receive irinotecan hydrochloride intravenously (IV) over 90 minutes on day 1 and oral erlotinib once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients per stratum receive escalating doses of erlotinib hydrochloride and irinotecan hydrochloride until the MTD is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Additional patients are treated at the MTD.

Patients are followed for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy that overexpresses epidermal growth factor receptor (EGFR)
* Unresectable disease for which there is no known standard therapy that ispotentially curative or definitely capable of extending life expectancy
* UGT1A1 genotype 6/6, 6/7, or 7/7
* Willing to provide biologic specimens
* Lesions amenable for 2 biopsies from the same tumor site (only patients receiving MTD in groups 2 and 3)
* No known brain metastases
* Performance status - ECOG 0-2
* At least 12 weeks
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST ≤ 2.5 times ULN (5 times ULN if liver metastases present)
* Creatinine no greater than 1.5 times ULN
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No New York Heart Association class III or IV heart disease
* No gastrointestinal tract disease resulting in an inability to take oral or nasogastric medication
* No requirement for IV alimentation
* No active peptic ulcer disease
* No abnormalities of the cornea (e.g., dry eye syndrome or Sjögren's syndrome)
* No congenital abnormality (e.g., Fuch's dystrophy)
* No abnormal slit-lamp examination using a vital dye (e.g., fluorescein or Bengal-Rose)
* No abnormal corneal sensitivity test (e.g., Schirmer test or similar tear production test)
* No other uncontrolled concurrent illness
* No ongoing or active infection
* No significant traumatic injury within the past 21 days
* No seizure disorder
* No psychiatric illness or social situation that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent grapefruit or grapefruit juice
* No smoking during study
* More than 4 weeks since prior immunotherapy or biologic therapy
* No concurrent immunotherapy
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No other concurrent chemotherapy
* Not specified
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to more than 25% of bone marrow
* No concurrent radiotherapy
* More than 3 weeks since prior major surgery
* No prior surgical procedures affecting absorption
* No prior EGFR-targeting therapy (e.g., gefitinib or EKB-569)
* No other concurrent investigational therapy
* No concurrent enzyme-inducing anticonvulsants (e.g., phenytoin, phenobarbital, carbamazepine, or valproic acid)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent enrollment on another study involving pharmacological agents for symptom control or therapeutic intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-06-13 (Actual); Primary Completion 2013-09-13 (Actual); Study Completion 2026-08-22 (Estimated)

PRIMARY OUTCOMES:
MTD of erlotinib hydrochloride and irinotecan hydrochloride in patients with advanced solid tumors that overexpress epidermal growth factor receptor | At least 4 weeks
  Defined as the highest safely tolerated dose where at most one patient experiences DLT with the next higher dose having at least 2 patients who experience DLT. Three patients will be entered at a given dose level and observed for at least 4 weeks to assess toxicity. MTD will be determined independently for each cohort.
Dose limiting toxicity of the combination in all cohorts | At least 4 weeks
  Defined as an adverse event attributed (definitely, probably, or possibly) to the study treatment. Graded using the National Cancer Institute Common Toxicity Criteria (CTC) version 2.0. Defined by the NCI Common Terminology Criteria for Adverse Events (CTCAE) versioun 4.0.
Effect of erlotinib hydrochloride on the disposition of irinotecan hydrochloride | Weekly during course 1
  Analysis performed using high performance liquid chromatography assays. Serial blood samples will be obtained during Cycle 1 only to determine the pharmacokinetics of irinotecan hydrochloride and erlotinib hydrochloride.
Effect of erlotinib on EGFR phosphorylation at MTD | Weekly during course 1
Genetic variation in UGT1A1 and BCRP | Weekly during course 1
  Detected using allele-specific restriction fragment length polymorphism (RFLP) assays and GeneScan assays. The overall incidence of UTG1A1 polymorphism will be estimated and summarized.
Tumor BCRP expression in patients treated at the MTD | Weekly during course 1
Evidence of anti tumor activity | Every 3 weeks
  Evaluated using modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
Correlation of EGFR phosphorylation and/or BCRP expression with response to this combination | Every 3 weeks
  Evaluated using modified RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Henry C Pitot, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States